CLINICAL TRIAL: NCT04678960
Title: Preventing Opioid Use Among Justice-involved Youth as They Transition to Adulthood: Leveraging Safe Adults (LeSA)
Brief Title: Preventing Opioid Use Among Justice-involved Youth as They Transition to Adulthood Leveraging Safe Adults (LeSA)
Acronym: LeSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UH3DA050250 (NIH)
Record Dates: First submitted 2020-11-11; First posted 2020-12-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use; Substance Use
Keywords: trauma-informed care; justice-involved youth; prevention for opioid use and other substances; Trust-based relational intervention (TBRI); youth-caregiver relationship
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: An effectiveness-Implementation Hybrid Design - Type 1; Randomized controlled trial and delayed-start study testing the effectiveness of Trust-based Relational Intervention and three different support formats (no coaching/structured coaching/adaptive coaching) among Juvenile Justice (JJ)-involved youth transitioning to their communities and a safe adult (e.g. parent/guardian, extended family member). In the delayed-start design, JJ agencies are randomly assigned to four different starting points with two months apart for starting the project. The last 18-months of the delayed-start design will provide a naturalistic investigation of sustainment of the intervention within the facilities after responsibility for intervention delivery has been transferred from TCU to the JJ agencies (TCU provide trainings to foster in-house TBRI expertise and assistance for implementation).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Reentry Practice (No Intervention): Youth/safe adult participants only receive assessments (baseline assessment while youth are at the facility; 3, 6, 12, 18 months follow-up assessments after youth are released from the facility).
- TBRI Training only (Experimental): Youth/safe adult dyads participate in 9 TBRI caregiver modules (caregivers only), 9 youth modules (youth only), and 4 Nurture Groups (caregiver and youth joint role-play activities) prior to youth's release.
  After the youth's release, they would receive phone support (only when requested by the caregiver or youth).
  Interventions: Behavioral: Trust-based Relational Intervention Training
- TBRI Training + TBRI In-Home Structured Coaching (Experimental): Youth/safe adult dyads participate in 9 TBRI caregiver modules (caregivers only), 9 youth modules (youth only), and 4 Nurture Groups (caregiver and youth joint role-play activities) prior to youth's release.
  After youth's release, trained TCU TBRI Practitioners provide coaching sessions to youth/safe adult dyads in which they meet 4 times (once monthly) over the first 4 months following release.
  Interventions: Behavioral: Trust-based Relational Intervention Training; Behavioral: Trust-based Relational Intervention In-Home Structured Coaching
- TBRI Training + TBRI In-Home Responsive Coaching (Experimental): Youth/safe adult dyads participate in 9 TBRI caregiver modules (caregivers only), 9 youth modules (youth only), and 4 Nurture Groups (caregiver and youth joint role-play activities) prior to youth's release.
  After youth's release, trained TCU TBRI Practitioners provide coaching sessions to youth/safe adult dyads. They meet a minimum of 2 times during the first 2 months after release. Starting from Month 3, TBRI Practitioners would provide additional coaching when requested or when a research assistant (RA) identifies a need for additional coaching sessions.
  Interventions: Behavioral: Trust-based Relational Intervention Training; Behavioral: Trust-based Relational Intervention In-Home Responsive Coaching

INTERVENTIONS:
Behavioral: Trust-based Relational Intervention Training — The intervention (Trust-based Relational Intervention® TBRI®) uses a youth-centered, attachment-based, and trauma-informed approach to strengthen youth/safe adult relationships and improve youth self-regulation (thinking, emotions, and behavior). TBRI includes TBRI Group Training and TBRI In-Home Coaching.
  TBRI Group Training is comprised of three components: TBRI Youth Group Training (youth only), Caregiver Training (caregivers only), and Nurture Groups (youth-caregiver joint roleplay activities), which is conducted prior to youth's release.
  Other Names: TBRI
  Arms: TBRI Training + TBRI In-Home Responsive Coaching; TBRI Training + TBRI In-Home Structured Coaching; TBRI Training only
Behavioral: Trust-based Relational Intervention In-Home Structured Coaching — The intervention (Trust-based Relational Intervention® TBRI®) uses a youth-centered, attachment-based, and trauma-informed approach to strengthen youth/safe adult relationships and improve youth self-regulation (thinking, emotions, and behavior). TBRI includes TBRI Group Training and TBRI In-Home Coaching.
  TBRI In-Home Structured Training includes four structured in-home coaching sessions.
  Other Names: TBRI Structured Coaching
  Arms: TBRI Training + TBRI In-Home Structured Coaching
Behavioral: Trust-based Relational Intervention In-Home Responsive Coaching — The intervention (Trust-based Relational Intervention® TBRI®) uses a youth-centered, attachment-based, and trauma-informed approach to strengthen youth/safe adult relationships and improve youth self-regulation (thinking, emotions, and behavior). TBRI includes TBRI Group Training and TBRI In-Home Coaching.
  TBRI In-Home Responsive Training includes at least 2 structured in-home coaching sessions plus additional sessions indefinitely as needed.
  Other Names: TBRI Responsive Coaching
  Arms: TBRI Training + TBRI In-Home Responsive Coaching

SUMMARY:
Across the US, substance use is a significant public health concern, with juvenile justice (JJ)-involved youth representing a particularly vulnerable population. The current study proposes to adapt and test an intervention Trust-based Relational Intervention® (TBRI®) for preventing initiation and/or escalation of opioid misuse among older adolescents involved in the JJ system. Successful completion of study aims will provide information on TBRI's utility for older JJ adolescents, barriers and facilitators of sustainment, and provide training and implementation support for sustainment in participating facilities.

DETAILED DESCRIPTION:
Across the US, substance use (SU) is a significant public health concern, with an estimated 11.1 million misusing prescription opioids. Rates of opioid use disorders (OUDs) have increased exponentially, with 60% of overdoses attributed to heroin and illicit synthetics (such as Fentanyl). Although opioid use among youth is low compared to adults, experimentation and regular use increases later in adolescence as youth transition to adulthood. Juvenile justice (JJ)-involved youth represent a particularly vulnerable population, as they often experience mental health disorders, dysfunctional family/social relationships, and complex trauma, placing them at greater risk for SU and substance use disorders (SUDs). To ensure that these youth do not become another opioid statistic, innovative and effective prevention interventions are needed. The investigators propose to adapt and test an intervention for preventing initiation and/or escalation of opioid misuse among older JJ-involved adolescents. The target enrollment group will be youth aging out of JJ (15-18 years at study enrollment) who are transitioning to their communities after a period of detainment in a secure treatment or correctional facility. Trust-based Relational Intervention® (TBRI®; a relational, attachment-based intervention that promotes emotional regulation through interaction with responsive adults) will be adapted as a prevention intervention targeting youth at risk for SU (especially non-medical use of opioids). Safe adults (e.g., parent/guardian, extended family member) will be trained in behavior management techniques for empowering youth to appropriately express their needs, connecting them with others in pro-social ways, and correcting or reshaping undesirable behavior. The proposed Effectiveness/Implementation study will examine both the effectiveness of TBRI for preventing opioid misuse and the comparative utility of three support formats: (1) TBRI Training only, (2) TBRI Training + Structured Coaching, or (3) TBRI Training + Responsive Coaching (triggered by the youth's need/risk). A total of 360 youth/safe adult dyads will be recruited from 9 participating JJ facilities over a 3-year period, and followed for 18 months post-release (15 youth-adult dyads/year per facility). This design enables a comparison of TBRI versus Standard Reentry Practice (SRP; using a stepped-wedge design where each facility serves as its own control) plus a randomized control trial comparing 3 TBRI support formats. This study will also examine barriers and facilitators of TBRI sustainment. Ninety JJ staff (10 from each agency) will provide input annually via focus groups and surveys. TCU will work with administrators and staff at each JJ facility to implement a sustainment plan, which will include developing in-house TBRI expertise (i.e., staff training and implementation assistance). Successful completion of study aims will provide a test of the adapted intervention and will facilitate sustainment by providing training and implementation support to participating facilities.

ELIGIBILITY:
Inclusion Criteria:

For the effectiveness component,

* Youth ages 15-18 at study enrollment
* Being disposed to community supervision (i.e., probation) following a minimum of 2 months in the secure residential JJ facility
* No indication of active suicide risk
* Being able to identify one safe adult that is willing to participate in the study.

For the implementation component:

• All staff with direct care or supervisory responsibilities within and outside the facilities (i.e., officers supervising youth after release) working with TCU on the LeSA project.

Exclusion Criteria:

* Youth outside the age range described above
* Active suicide risk at the time of recruitment

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Youth days to opioid (and other substance use) initiation | 15 months
  Initiation to opioid and other substance use (e.g., alcohol, marijuana, methamphetamine) over 15 months follow-up in days, measured by the scale of Timeline follow-back, Substance Use Involvement (i.e., during the past 30 days, how many days did you use alcohol or drugs; developed by the HEAL Prevention Cooperative), urinalysis results. Scores: 0-450 days; a higher score indicating a better outcome.
Youth months to opioid (and other substance use) initiation | 15 months
  Initiation to opioid and other substance use over 15 months follow-up in months, monthly check-ins (any opioid use; any alcohol, other drug use in the past month). Scores: 0-15 months; a higher score indicating a better outcome.
Youth substance use severity | 15 months
  Opioid use and other substance use (e.g., alcohol, marijuana, methamphetamine) over 15 months; measured by TCU Drug Screen 5 and TCU Drug Screen 5 - Opioid Supplement. Scores: 0-11, a higher score indicating a worse outcome.

SECONDARY OUTCOMES:
Self-regulation (youth) - positive and negative urgency | 15 months
  TCU Adolescent Thinking Forms (TCU THK); Scores: 10-50; a higher score indicating a worse outcome
Self-regulation (youth) - delayed discounting | 15 months
  Delay Discounting Task; Scores: 1-13; a higher score indicating a better outcome
Self-regulation (youth) - emotion regulation | 15 months
  Difficulties in Emotion Regulation. Scores: 1-5, a higher score indicating a worse outcome
Self-regulation (youth) - executive functioning | 15 months
  Barkley Deficits in Executive Functioning Scale-Child and Adolescent Short Form. Scores: 1-4, a higher score indicating a worse outcome.
Self-efficacy (youth) | 15 months
  Two items (developed by the HEAL Prevention Cooperative) assessing how confident participants not misuse prescription or heroin in the next 30 days. Scores: 0-4, a higher score indicating a better outcome
Social exposure to alcohol, marijuana, heroin, and prescription opioids (youth) | 15 months
  Four items, developed by the HEAL Prevention Cooperative, to assess social exposure to alcohol, marijuana, heroin, and prescription opioids (i.e., how often the adult who is most important to the participant drink alcohol or use marijuana, heroin, and prescription opioids). Scores: 0-3, a higher score indicating a worse outcome
Behavioral problems (youth) | 15 months
  Behavioral problems in the areas of peer problems, hyperactivity, emotional problems, and conduct problems, assessed by the Strength and Difficulties Questionnaire. Scores: 0-40, a higher score indicating a worse outcome
Prosocial behavior (youth) | 15 months
  Prosocial behavior is assessed by the Prosocial subscale of the Strength and Difficulties Questionnaire. Scores: 0-10, a higher score indicating a better outcome.
Monthly check-ins on behavioral misconduct (youth) | 15 months
  Monthly check-ins asking any truancy, trouble with the law during the last month. Scores: 0 (no) or 1 (yes, being involved in the behavioral misconduct).
Anxiety (both youth and caregivers) | 15 months
  Assessed by the General Anxiety Disorder (GAD) -7. Scores: 0-3, a higher score indicating a worse outcome.
Depression (both youth and caregivers) | 15 months
  Assessed by the Patient Health Questionnaire (PHQ). Scores: 0-3, a higher score indicating a worse outcome.
Pain (both youth and caregivers) | 15 months
  Assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain domain. Scores: 0-3, a higher score indicating a worse outcome.
Youth and caregiver relationship | 15 months
  Assessed by the Experiences in Close Relationships. Scores: 1-7, a higher score indicating a worse outcome.
Family relationship | 15 months
  Assessed by the Family Assessment Device. Scores: 1-4, a higher score indicating a better outcome.
Monthly check-ins on anxiety, depression, and stress in the relationship with caregiver/safe adult (youth) | 15 months
  Monthly check-ins asking any increase in anxiety, depression, or stress in the relationship with caregiver/safe adult. Scores: 0 (no) or 1 (yes, there is an increase in the past month).

OTHER OUTCOMES:
Frequency of receiving substance use treatment | 15 months
  Frequency of receiving substance use treatment (alcohol, illegal drug use). Scores: 0 (never), 1 (once), or 2 (more than once), a higher score indicating a worse outcome.
Times of hospital visits related to substance use | 15 months
  Times of hospital visits related to substance use. Scores: 0 - the number of times. A higher score indicating a worse outcome.
Times of treatment referral for substance use | 15 months
  Times of treatment referral for substance use. Scores: 0 - the number of times. A higher score indicating a worse outcome.
Frequency of opioid overdose | 15 months
  Frequency of opioid overdose. Scores: 0 (never), 1 (once), or 2 (more than once), a higher score indicating a worse outcome.
Receipt of Narcan for opioid overdose | 15 months
  Receipt of Narcan for opioid overdose. Scores: 0 (no) or 1 (yes), a score of 1 indicating a worse outcome.
Recidivism | 15 months
  Whether or not youth are re-arrest (0 = no, 1 = yes) or re-adjudicated (0 = no, 1 = yes). The information will come from JJ agency youth records. A score of 1 indicating a worse outcome.
Recidivism | 15 months
  Days between discharge and youth's re-arrest and re-adjudication. The information will come from JJ agency youth records. Scores: 0-450 days, a higher score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Danica K Knight, Ph.D., Principal Investigator — Texas Christian University
Locations (11):
- United States (11):
  - Illinois Youth Center - Chicago, Chicago, Illinois
  - Illinois Youth Center - Pere Marquette, Grafton, Illinois
  - Illinois Youth Center- Harrisburg, Harrisburg, Illinois
  - Illinois Youth Center- Warrenville, Naperville, Illinois
  - Illinois Youth Center - St. Charles, St. Charles, Illinois
  - Grayson County Juvenile Center/Boot Camp, Denison, Texas
  - Texas Monarch Academy for Girls/Rite of Passage, Denison, Texas
  - Williamson County Juvenile Services, Georgetown, Texas
  - Lake Granbury Youth Services/Rite of Passage, Granbury, Texas
  - Harris County Youth Village, Houston, Texas
  - Collin County Juvenile Probation Services, McKinney, Texas

IPD SHARING:
Plan to Share IPD: Yes
All data will be further de-identified (e.g., by systematically scrambling Study IDs within study sites) before being shared with the HEAL Prevention Coordinating Center. The Coordinating Center will not have access to identifying information, nor will they have access to or knowledge of how participant study identification numbers were scrambled.
  The data will also be shared publicly, following the HEAL Prevention Guidance for Appropriate Public Access and Data Sharing Plans, including the following aspects:
  * Electronic copies of publications will be deposited within 4 weeks of acceptance
  * Publications will be published under the Creative Commons Generic License
  * Publications will be made publicly available immediately without embargo
  * Underlying Primary Data for the Publications will be made broadly available
  * Sharing of Underlying Primary Data must be responsive to protecting confidential and proprietary data and is consistent with applicable laws and regulations.
Time Frame: The data will be shared with the HEAL Prevention Cooperative between 2021 and 2024.
  Sharing of underlying primary data for the publications will be made broadly available through an appropriate data repository, such as the NIH HEAL Initiative central data repository, or a non-NIH repository that conforms to the principles articulated in the HEAL Public Access and Data Sharing Policy (referred to in the URL included below).
Access Criteria: All research teams that participate in the NIH Helping to End Addiction Long-term (HEAL) Initiative.
  https://heal.nih.gov/files/2020-01/2020-01-16_data-sharing-4.pdf
URL: https://heal.nih.gov/about/public-access-data

REFERENCES:
- [Background] Biederman J, Faraone SV, Monuteaux MC, Feighner JA. Patterns of alcohol and drug use in adolescents can be predicted by parental substance use disorders. Pediatrics. 2000 Oct;106(4):792-7. doi: 10.1542/peds.106.4.792. PMID 11015524
- [Background] Baglivio, M. T., & Epps, N. (2016). The interrelatedness of adverse childhood experiences among high-risk juvenile offenders. Youth Violence and Juvenile Justice, 14(3), 179-198.
- [Background] Baglivio, M. T., Wolff, K. T., Piquero, A. R., & Epps, N. (2015). The relationship between Adverse Childhood Experiences (ACE) and juvenile offending trajectories in a juvenile offender sample. Journal of Criminal Justice, 43(3), 229-241.
- [Background] Belenko S, Johnson ID, Taxman FS, Rieckmann T. Probation Staff Attitudes Toward Substance Abuse Treatment and Evidence-Based Practices. Int J Offender Ther Comp Criminol. 2018 Feb;62(2):313-333. doi: 10.1177/0306624X16650679. Epub 2016 May 23. PMID 27220361
- [Background] Brockie TN, Dana-Sacco G, Wallen GR, Wilcox HC, Campbell JC. The Relationship of Adverse Childhood Experiences to PTSD, Depression, Poly-Drug Use and Suicide Attempt in Reservation-Based Native American Adolescents and Young Adults. Am J Community Psychol. 2015 Jun;55(3-4):411-21. doi: 10.1007/s10464-015-9721-3. PMID 25893815
- [Background] Brown LK, Tarantino N, Tolou-Shams M, Esposito-Smythers C, Healy MG, Craker L. Mental Health Symptoms and Parenting Stress of Parents of Court-Involved Youth. J Child Fam Stud. 2018 Mar;27(3):843-852. doi: 10.1007/s10826-017-0923-1. Epub 2017 Nov 6. PMID 29805245
- [Background] Colder CR, Shyhalla K, Frndak SE. Early alcohol use with parental permission: Psychosocial characteristics and drinking in late adolescence. Addict Behav. 2018 Jan;76:82-87. doi: 10.1016/j.addbeh.2017.07.030. Epub 2017 Jul 25. PMID 28772246
- [Background] Council of State Governments Justice Center. (2017, September). Dos and don'ts for reducing recidivism among young adults in the justice system. Retrieved February 15, 2019 from https://csgjusticecenter.org/wp-content/uploads/2017/09/Dos-and-Donts-for-Reducing- Recidivism-among-Young-Adults-in-the-Justice-System.pdf
- [Background] Dube SR, Miller JW, Brown DW, Giles WH, Felitti VJ, Dong M, Anda RF. Adverse childhood experiences and the association with ever using alcohol and initiating alcohol use during adolescence. J Adolesc Health. 2006 Apr;38(4):444.e1-10. doi: 10.1016/j.jadohealth.2005.06.006. PMID 16549308
- [Background] Evans-Chase, M. (2014). Addressing trauma and psychosocial development in juvenile justice- involved youth: A synthesis of the developmental neuroscience, juvenile justice and trauma literature. Laws, 3(4), 744-758. DOI: 10.3390/laws3040744
- [Background] Ford, J. D., & Hawke, J. (2012). Trauma affect regulation psychoeducation group and milieu intervention outcomes in juvenile detention facilities. Journal of Aggression, Maltreatment & Trauma, 21(4), 365-384. https://doi.org/10.1080/10926771.2012.673538
- [Background] Forster M, Grigsby TJ, Rogers CJ, Benjamin SM. The relationship between family-based adverse childhood experiences and substance use behaviors among a diverse sample of college students. Addict Behav. 2018 Jan;76:298-304. doi: 10.1016/j.addbeh.2017.08.037. Epub 2017 Sep 1. PMID 28889058
- [Background] Fosco GM, Frank JL, Stormshak EA, Dishion TJ. Opening the "Black Box": family check-up intervention effects on self-regulation that prevents growth in problem behavior and substance use. J Sch Psychol. 2013 Aug;51(4):455-68. doi: 10.1016/j.jsp.2013.02.001. Epub 2013 Feb 26. PMID 23870441
- [Background] Frisman, L., Ford, J., Lin, H.-J., Mallon, S., & Chang, R. (2008). Outcomes of trauma treatment using the TARGET Model. https://doi.org/10.1080/15560350802424910
- [Background] Hovdestad, W. E., Tonmyr, L., Wekerle, C., & Thornton, T. (2011). Why is childhood maltreatment associated with adolescent substance abuse? A critical review of explanatory models. International Journal of Mental Health Addiction, 9(5), 525-542. DOI: 10.1007/s11469-011-9322-9
- [Background] Kumpfer KL, Alvarado R, Whiteside HO. Family-based interventions for substance use and misuse prevention. Subst Use Misuse. 2003 Sep-Nov;38(11-13):1759-87. doi: 10.1081/ja-120024240. PMID 14582577
- [Background] Laird RD, Pettit GS, Bates JE, Dodge KA. Parents' monitoring-relevant knowledge and adolescents' delinquent behavior: evidence of correlated developmental changes and reciprocal influences. Child Dev. 2003 May-Jun;74(3):752-68. doi: 10.1111/1467-8624.00566. PMID 12795388
- [Background] Marrow, M. T., Knudsen, K. J., Olafson, E., & Bucher, S. E. (2012). The value of implementing TARGET within a trauma-informed Juvenile Justice Setting. Journal of Child & Adolescent Trauma, 5(3), 257-270. DOI: 10.1080/19361521.2012.697105
- [Background] Murray, D. W., Rosanbalm, K., & Christopoulos, C. (2016, February). Self-Regulation and toxic stress report 3: A comprehensive review of self-regulation interventions from birth through young adulthood (OPRE Report # 2016-34). Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services. Retrieved February 14, 2019 from https://www.acf.hhs.gov/sites/default/files/opre/acf_report_3_approved_fromword_b508. pdf
- [Background] National Center for Mental Health and Juvenile Justice. (2016, September). Trauma among youth in the Juvenile Justice System. Retrieved March 7, 2019 from https://www.ncmhjj.com/wp-content/uploads/2016/09/Trauma-Among-Youth-in-the- Juvenile-Justice-System-for-WEBSITE.pdf
- [Background] Nelis D, Kotsou I, Quoidbach J, Hansenne M, Weytens F, Dupuis P, Mikolajczak M. Increasing emotional competence improves psychological and physical well-being, social relationships, and employability. Emotion. 2011 Apr;11(2):354-66. doi: 10.1037/a0021554. PMID 21500904
- [Background] National Research Council (US) and Institute of Medicine (US) Committee on the Prevention of Mental Disorders and Substance Abuse Among Children, Youth, and Young Adults: Research Advances and Promising Interventions; O'Connell ME, Boat T, Warner KE, editors. Preventing Mental, Emotional, and Behavioral Disorders Among Young People: Progress and Possibilities. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK32775/ PMID 20662125
- [Background] Quinn K, Frueh BC, Scheidell J, Schatz D, Scanlon F, Khan MR. Internalizing and externalizing factors on the pathway from adverse experiences in childhood to non-medical prescription opioid use in adulthood. Drug Alcohol Depend. 2019 Apr 1;197:212-219. doi: 10.1016/j.drugalcdep.2018.12.029. Epub 2019 Feb 14. PMID 30849646
- [Background] Robertson AA, Xu X, Stripling A. Adverse events and substance use among female adolescent offenders: effects of coping and family support. Subst Use Misuse. 2010 Feb;45(3):451-72. doi: 10.3109/10826080903452512. PMID 20141458
- [Background] Shin SH, McDonald SE, Conley D. Patterns of adverse childhood experiences and substance use among young adults: A latent class analysis. Addict Behav. 2018 Mar;78:187-192. doi: 10.1016/j.addbeh.2017.11.020. Epub 2017 Nov 13. PMID 29179155
- [Background] Stein MD, Conti MT, Kenney S, Anderson BJ, Flori JN, Risi MM, Bailey GL. Adverse childhood experience effects on opioid use initiation, injection drug use, and overdose among persons with opioid use disorder. Drug Alcohol Depend. 2017 Oct 1;179:325-329. doi: 10.1016/j.drugalcdep.2017.07.007. Epub 2017 Aug 5. PMID 28841495
- [Background] Steinberg L. Risk taking in adolescence: what changes, and why? Ann N Y Acad Sci. 2004 Jun;1021:51-8. doi: 10.1196/annals.1308.005. PMID 15251873
- [Background] Taxman FS, Young DW, Fletcher BW. The National Criminal Justice Treatment Practices survey: an overview of the special issue. J Subst Abuse Treat. 2007 Apr;32(3):221-3. doi: 10.1016/j.jsat.2006.12.017. Epub 2007 Mar 9. No abstract available. PMID 17383547
- [Background] Texas Senate Bill 1356. (2013, September 1). About Texas Senate Bill 1356. Retrieved March 8, 2019 from https://www.crisisprevention.com/Blog/August-2013/Texas-Senate-Bill-1356?lang=en-US
- [Background] Tolou-Shams M, Brogan L, Esposito-Smythers C, Healy MG, Lowery A, Craker L, Brown LK. The role of family functioning in parenting practices of court-involved youth. J Adolesc. 2018 Feb;63:165-174. doi: 10.1016/j.adolescence.2017.12.016. Epub 2018 Jan 6. PMID 29310009
- [Background] Tolou-Shams M, Hadley W, Conrad SM, Brown LK. The Role of Family Affect in Juvenile Drug Court Offenders' Substance Use and HIV Risk. J Child Fam Stud. 2012 Jun 1;21(3):449-456. doi: 10.1007/s10826-011-9498-4. Epub 2011 May 6. PMID 22661883
- [Background] Wills, T. A., Sandy, J. M., Shinar, O., & Yaeger, A. (1999). Contributions of positive and negative affect to adolescent substance use: Test of a bidimensional model in a longitudinal study. Psychology of Addictive Behaviors, 13(4), 327-338. http://dx.doi.org/10.1037/0893-164X.13.4.327
- [Background] Wills TA, Sandy JM, Yaeger AM. Moderators of the relation between substance use level and problems: test of a self-regulation model in middle adolescence. J Abnorm Psychol. 2002 Feb;111(1):3-21. PMID 11866177
- [Background] Wolff KT, Baglivio MT, Piquero AR. The Relationship Between Adverse Childhood Experiences and Recidivism in a Sample of Juvenile Offenders in Community-Based Treatment. Int J Offender Ther Comp Criminol. 2017 Aug;61(11):1210-1242. doi: 10.1177/0306624X15613992. Epub 2015 Nov 12. PMID 26567183
- [Background] Wright, K. N., & Wright, K. E. (1993). Family life and delinquency and crime: A policymakers' guide to the literature (NCJ 140517). Washington, DC: U.S. Department of Justice, Office of Juvenile Justice and Delinquency Prevention, National Institute of Justice. Retrieved March 8, 2019 from https://www.ncjrs.gov/pdffiles1/Digitization/140517NCJRS.pdf
- [Background] Zolkoski, S. M., & Bullock, L. M. (2012). Resilience in children and youth: A review. Children and Youth Services Review, 34(12), 2295-2303. http://dx.doi.org/10.1016/j.childyouth.2012.08.009
- [Derived] Kuklinski MR, Gibbons BJ, Bowser DM, McCollister KE, Smart R, Dunlap LJ, Shenkar E, Bonar EE, Boomer T, Campbell M, Fiellin LE, Hutton DW, Rao V, Saldana L, Su K, Walton MA, Yilmazer T. Investing in Interventions to Prevent Opioid Use Disorder in Adolescents and Young Adults: Start-up Costs from NIDA's HEAL Prevention Initiative. Prev Sci. 2025 Nov;26(7):1045-1055. doi: 10.1007/s11121-025-01835-6. Epub 2025 Oct 14. PMID 41085955
- [Derived] Bowser D, McCollister K, Berchtold G, Ruscitti B, Yang Y, Hines H, Fardone E, Knight D. Start-Up and Implementation Costs for the Trust Based Relational Intervention. J Prev (2022). 2024 Dec;45(6):847-860. doi: 10.1007/s10935-024-00803-0. Epub 2024 Aug 17. PMID 39153158
- [Derived] Razuri EB, Yang Y, Tinius E, Knight DK. Adaptation of a trauma-informed intervention to prevent opioid use among youth in the legal system. J Subst Use Addict Treat. 2024 Aug;163:209294. doi: 10.1016/j.josat.2024.209294. Epub 2024 Jan 24. PMID 38272116
- [Derived] Ahrens K, Blackburn N, Aalsma M, Haggerty K, Kelleher K, Knight DK, Joseph E, Mulford C, Ryle T, Tolou-Shams M. Prevention of Opioid Use and Disorder Among Youth Involved in the Legal System: Innovation and Implementation of Four Studies Funded by the NIDA HEAL Initiative. Prev Sci. 2023 Oct;24(Suppl 1):99-110. doi: 10.1007/s11121-023-01566-6. Epub 2023 Jul 1. PMID 37393415
- [Derived] Razuri EB, Yang Y, Tinius E, Knight DK. Adaptation of a trauma-informed intervention for youth involved in the legal system. Res Sq [Preprint]. 2023 Mar 1:rs.3.rs-2596631. doi: 10.21203/rs.3.rs-2596631/v1. PMID 36909596
- [Derived] Knight DK, Yang Y, Joseph ED, Tinius E, Young S, Shelley LT, Cross DR, Knight K. Preventing opioid use among justice-involved youth as they transition to adulthood: leveraging safe adults (LeSA). BMC Public Health. 2021 Nov 20;21(1):2133. doi: 10.1186/s12889-021-12127-3. PMID 34801009